CLINICAL TRIAL: NCT03707184
Title: [18F]Fluciclovine Companion Imaging Study to Radium-223 and Radiotherapy in Hormone-Naive Men With Oligometastatic Prostate Cancer to Bone (RROPE) Study
Brief Title: Fluciclovine F18 PET/CT Imaging in Assessing Hormone-Naive Men With Prostate Cancer That Has Spread to the Bone
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HCI113970; NCI-2018-02083 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2018-10-09; First posted 2018-10-16 (Actual); Results first posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Metastatic Prostate Carcinoma; Prostate Carcinoma Metastatic in the Bone; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — fluciclovine F-18; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic (fluciclovine F18, PET/CT) (Experimental): Patients receive fluciclovine F18 intravenously (IV) over 30 seconds and undergo PET/CT scan over 60 minutes at baseline, 3 months and at approximately 6 months of radium-223 therapy.
  Interventions: Procedure: Computed Tomography; Drug: Fluciclovine F18; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo PET/CT scan
  Other Names: CAT; CAT Scan; Computerized Axial Tomography (CAT); computerized tomography; CT; CT Scan; tomography
Drug: Fluciclovine F18 — Given IV
  Other Names: (18F)Fluciclovine; 18F-Fluciclovine; Fluciclovine (18F)
Procedure: Positron Emission Tomography — Undergo PET/CT scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This trial studies how well fluciclovine 18F PET/CT imaging works in assessing hormone-naive men with prostate cancer that has spread to the bone. Fluciclovine 18F is a radioactive drug used to measure tumor growth. PET/CT uses x-rays to take pictures inside the body. Comparing results of fluciclovine 18F PET/CT imaging may help doctors predict a patient's response to treatment and help plan the best treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Abnormal fluciclovine F18 ([18F] fluciclovine) uptake on visual assessment will differ by the type of metastatic lesion present (blastic, lytic, marrow, mixed).

II. Maximum standardized uptake value (SUVmax) and mean standardized uptake value (SUVmean) on (18F) fluciclovine-positron emission tomography (PET)/computed tomography (CT) imaging will differ by the type of metastatic lesion present (blastic, lytic, marrow, mixed).

SECONDARY OBJECTIVES:

I. Determine if a 25% or greater reduction in average (ave) SUVmax or ave SUVmean on (18F) fluciclovine-PET/CT imaging after completion of all radiation therapy will be predictive of increased time to biochemical failure.

II. Determine the correlation between the number of lesions, their visual uptake, and semi-quantitative uptake on technetium tc-99m medronate (99mTc-MDP) bone scintigraphy and (18F) fluciclovine- PET/CT at baseline.

III. Determine the correlation between the number of lesions, their visual uptake, and semi-quantitative uptake on 99mTc-MDP bone scintigraphy and (18F) fluciclovine- PET/CT after 3 and 6 cycles of treatment.

OUTLINE: This is a companion imaging study to Institutional Review Board (IRB) #102312 (A Phase 2 Study of Radium-223 and Radiotherapy in Hormone-Naive Men with Oligometastatic Prostate Cancer to Bone).

Patients receive fluciclovine F18 intravenously (IV) over 30 seconds and undergo PET/CT scan over 60 minutes at baseline, 3 months and at approximately 6 months of radium-223 therapy.

After completion of diagnostic testing, patients are followed for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment on IRB #102312 (A Phase 2 Study of Radium-223 and Radiotherapy in Hormone-Naive Men with Oligometastatic Prostate Cancer to Bone).
* Patients must document their willingness to be followed for up to 24 months after recruitment by signing informed consent documenting their agreement to allow access to the data obtained on IRB #102312 and information and data entered into a research database.
* All patients, or their legal guardians, must sign a written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization in accordance with institutional guidelines.

Exclusion Criteria:

* Patients with known allergic or hypersensitivity reactions to previously administered radiopharmaceuticals. Patients with significant drug or other allergies or autoimmune diseases may be enrolled at the Investigator?s discretion.
* Patients who require monitored anesthesia for PET scanning.
* Patients who are too claustrophobic to undergo PET scanning.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2022-02-03 (Actual); Study Completion 2022-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Yap, PhD, Principal Investigator — Huntsman Cancer Institute/ University of Utah
Locations (1):
- Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diagnostic (Fluciclovine F18, PET/CT)
Started | 17
Completed | 15
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Diagnostic (Fluciclovine F18, PET/CT)
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.41 (6.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Mean Standardized Uptake Value (SUVmean) by Lesion Type
Description: Mean SUV values are reported according to the type of bone lesion (osteoblastic dense, osteoblastic ground glass, osteoblastic mixed, and osteolytic).
Time Frame: Participants were assessed using [18F]Fluciclovine-PET/CT at baseline, prior to initiating radium-223 therapy
Population: The [18F]Fluciclovine-PET/CT scans were evaluated for 17 enrolled participants. The 19 lesions seen on PET that had a definitive CT correlate were categorized by lesion type. The number of units analyzed for each row reflect the number of lesions in each category. Some participants had multiple lesions of different types.
Measure: Mean (Standard Deviation); unit: SUV by body weight (kg)
Units Other Than Participants: Lesions
Groups:
- Diagnostic (Fluciclovine F18, PET/CT): Participants receive fluciclovine F18 intravenously (IV) over 30 seconds and undergo PET/CT scan over 60 minutes at baseline, 3 months and at approximately 6 months of radium-223 therapy.
  Computed Tomography: Undergo PET/CT scan
  Fluciclovine F18: Given IV
  Positron Emission Tomography: Undergo PET/CT scan
Arm/Group | Diagnostic (Fluciclovine F18, PET/CT)
Number analyzed (Participants) | 17
Number analyzed (Lesions) | 19
SUV by body weight (kg)
  Osteoblastic Dense | 1.91 (0.69)
  Osteoblastic Ground Glass: number analyzed (Lesions) | 13
  Osteoblastic Ground Glass | 2.36 (1.12)
  Osteoblastic Mixed: number analyzed (Lesions) | 11
  Osteoblastic Mixed | 2.63 (1.26)
  Osteolytic: number analyzed (Lesions) | 13
  Osteolytic | 3.05 (0.43)

2. Primary Outcome: Maximum Standardized Uptake Value (SUVmax) by Lesion Type
Description: Maximum SUV values are reported according to the type of bone lesion (osteoblastic dense, osteoblastic ground glass, osteoblastic mixed, and osteolytic).
Time Frame: Participants were assessed using [18F]Fluciclovine-PET/CT at baseline, prior to initiating radium-223 therapy
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SUV by body weight (kg)
Units Other Than Participants: lesions
Arm/Group | Diagnostic (Fluciclovine F18, PET/CT)
Number analyzed (Participants) | 17
Number analyzed (lesions) | 19
SUV by body weight (kg)
  Osteoblastic Dense | 4.80 (1.53)
  Osteoblastic Ground Glass: number analyzed (lesions) | 13
  Osteoblastic Ground Glass | 7.17 (3.75)
  Osteoblastic Mixed: number analyzed (Participants) | 6
  Osteoblastic Mixed: number analyzed (lesions) | 11
  Osteoblastic Mixed | 8.39 (5.61)
  Osteolytic: number analyzed (Participants) | 5
  Osteolytic: number analyzed (lesions) | 13
  Osteolytic | 10.02 (3.33)

ADVERSE EVENTS:
Time Frame: Adverse events were assessed for 24 hours following administration of [18F] Fluciclovine dose.
Description: The collection of any adverse events will begin when a patient receives their first dose of [18F] Fluciclovine and will end 24 hours after receiving that dose. As there is the potential for each patient to receive up to three scanning visits, each constituting a radioactive tracer to be injected into the mpatient, the adverse events will be monitored for 24 hours after each injection and subsequent scan.
Arm/Group | Diagnostic (Fluciclovine F18, PET/CT)
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-05): https://cdn.clinicaltrials.gov/large-docs/84/NCT03707184/Prot_SAP_000.pdf